CLINICAL TRIAL: NCT00997022
Title: Phase I Open-Label, Dose-Finding Study of BAY 43-9006 (Sorafenib) in High-risk Hepatocellular Cancer Patients After Liver Transplantation
Brief Title: Trial of Sorafenib in Hepatocellular Cancer (HCC) Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bayer (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD3519
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Hepatocellular Cancer
Keywords: HCC; High-risk Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Daily sorafenib taken orally
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Dose escalation:
  Dose level 1: 200mg of sorafenib daily
  Dose level 2: 200mg of sorafenib BID (twice daily)
  Dose level 3: 200mg QAM (taken every morning) and 400mg QPM (taken every evening)
  Dose level 4: 400mg BID (twice daily)
  Other Names: Nexavar

SUMMARY:
This Phase I study of sorafenib in high risk hepatocellular cancer patients after liver transplantation will study 24 subjects for about 5 years. Each subject will receive sorafenib for 6 months. Safety and effectiveness on the post transplant, high risk HCC patients will be studied.

DETAILED DESCRIPTION:
Sorafenib (BAY 43-9006) is an oral multi-kinase inhibitor with effects on tumor proliferation and angiogenesis. Sorafenib is approved for the treatment of patients with advanced renal cancer and unresectable hepatocellular carcinoma (HCC). The recommended daily dose of Sorafenib is 400 mg (2 x 200 mg tablets) taken twice daily without food (at least 1 hour before or 2 hours after a meal). Studies of single-agent sorafenib showed treatment was well-tolerated with manageable side effects. The results seen with sorafenib in the Phase III (SHARP) trial suggest that VEGF and RAF kinase inhibition prolong survival in patients with advanced HCC. It is not known whether a drug which is considered primarily cytostatic will be effective in preventing cancer recurrences in the setting of minimal residual disease.

This is a phase I, single center, open-label, dose-escalation study to determine the maximum tolerated dose (MTD) and overall safety profile of daily sorafenib as therapy to prevent HCC recurrence in liver transplant subjects with high-risk HCC. For each subject, the study will consist of two phases: a treatment phase and an extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* ECOG Performance Status 0-2
* Post liver transplant and have explants with histologically confirmed hepatocellular carcinoma.
* No evidence of HCC disease at study entry by imaging
* Eligible to start 4 weeks post transplant (29 days post transplant) as long as they are on stable doses of immunosuppressants.
* "High risk" for recurrence after transplantation
* Received prior surgical resection, chemoembolization or other local therapy prior to transplant.
* Have Child-Pugh Class A or compensated Child-Pugh Class B liver dysfunction at the start of therapy
* Have adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin ≥ 8.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 75,000/mm3
  * Total bilirubin ≤ 1.5 times ULN
  * ALT and AST ≤ 5 x ULN
  * Creatinine ≤ 1.5 times ULN
  * Albumin ≥ 2.5 mg/dl
* Women of childbearing potential must have a negative serum pregnancy test performed within 14 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Exhibit the ability to understand and willingness to sign a written informed consent regarding the study and alternative treatments.
* INR < 1.5 or a PT/PTT within normal limits.

Exclusion Criteria:

* Cardiac disease: Congestive heart failure > class II NYHA.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension, defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Active clinically serious infection > CTCAE Grade 2.
* Thromboembolic events such as a cerebrovascular accident (including transient ischemic attacks) within the past 6 months.
* Any hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture within 4 weeks of first dose of study drug.
* Evidence or history of bleeding diathesis or coagulopathy within 4 weeks of first dose of study drug.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin within 4 weeks of first dose of study drug.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Patients who are pregnant or breastfeeding. Breastfeeding should be discontinued if the patient is to be treated.
* Prior malignancy treated during the prior 5-years (other than localized non-melanoma carcinoma of the skin).
* Any condition or social situation that may limit patient's compliance with the study regimen
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis prior to enrollment.
* Known human immunodeficiency virus (HIV) infection (hepatitis B and hepatitis C infection will not be exclusion criteria.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any malabsorption problem which in the investigator's opinion would prevent adequate absorption of the sorafenib.
* On M-Tor inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of daily sorafenib | Every two weeks throughout six cycles

SECONDARY OUTCOMES:
Duration of disease free survival | Every three months for 2 years
Duration of progression free survival | Every three months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Abby Siegel, MD, MS, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Columbia University Medical Center, New York, New York